CLINICAL TRIAL: NCT04079465
Title: Automated Oxygen Control by O2matic to Patients Admitted With Acute Hypoxemia
Acronym: O2MATIC-ACUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Ejvind Frausing Hansen, Senior Consultant, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O2MATIC-ACUTE
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hypoxemic Respiratory Failure; Hypoxia; Hypoxemia; Respiratory Failure; Respiratory Insufficiency
Keywords: closed-loop; oxygen treatment
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O2matic (Active Comparator): Usual care plus O2matic controlled oxygen therapy for a maximum of 24 hours or until weaning from oxygen supplementation
  Interventions: Device: O2matic
- Manual (No Intervention): Usual care plus manual controlled oxygen therapy by nursing staff. O2matic is used in monitoring mode to measure SpO2 continuously.

INTERVENTIONS:
Device: O2matic — O2matic controls oxygen supply with a closed-loop feedback from a pulse oximeter. The aim is to maintain SpO2 within a predefined target interval according to guidelines for the specific condition causing hypoxemia, with the lowest possible supplementation of oxygen.
  Arms: O2matic

SUMMARY:
The aim of this study is to examine if automated oxygen delivery with O2matic allows for faster weaning from oxygen supply and better oxygen control than manually controlled oxygen therapy for patients admitted to the emergency department with acute hypoxemia. Furthermore it will be tested if O2matic compared to manual control allows for earlier discharge.

DETAILED DESCRIPTION:
Closed-loop control of oxygen therapy is described in the literature used for preterm infants, trauma patients, medical emergency use, and for patients with Chronic Obstructive Pulmonary Disease (COPD). O2matic is a closed-loop system that is based on continuous and non-invasive measurement of pulse rate and oxygen-saturation (SpO2). The algorithm in O2matic controls oxygen delivery with the aim of keeping the SpO2 within the desired interval, which could be 88-92 % for patients at risk of hypercapnia or 94-98 % for patients with pneumonia, asthma exacerbation, heart failure and other medical emergencies, according to guidelines from British Thoracic Society (BTS). SpO2-interval can be set for the individual patients, as can the range of acceptable oxygen-flow. If SpO2 or oxygen-flow cannot be maintained within the desired intervals an alarm will sound.

All studies on closed-loop systems have shown that this method is better than manually control by nurse to maintain saturation within the desired interval. Furthermore, some studies have indicated that closed-loop has the possibility to reduce admission time and to reduce time spent with oxygen therapy, due to more efficient and faster withdrawal from oxygen supplementation.

In the present study O2matic will be tested versus manual control, for patients admitted to the emergency department with acute hypoxemia due to any reason, except for carbon monoxide (CO) poisoning and other conditions where SpO2 is not a reliable measure of hypoxemia. During the study the patients will either have oxygen controlled with O2matic or manually by nursing staff for 24 hours or until discharge or weaning from oxygen supply. All patients will have continuous logging of pulse rate, oxygen-saturation and oxygen-flow with O2matic, but only in the O2matic active group, the algorithm will control oxygen-delivery.

The primary hypothesis is that O2matic compared to manual control allows for faster weaning from oxygen supplementation, and that more patients will be weaned from oxygen supplementation within a time frame of 24 hours. Furthermore it will be tested if O2matic compared to manual control allows for earlier hospital discharge. It will be tested if O2matic is better than manual control in maintaining oxygen-saturation within the desired interval and reducing time with unintended hypoxia and hyperoxia.

No safety issues has been reported in the literature. O2matic is approved in Europe with "Conformité Européenne" (CE) mark, and approved for clinical testing by The Danish Medicines Agency, The Ethics Committee in the Capital Region of Denmark and by the regional Data Protection Board. The study will be conducted according to Good Clinical Practice (GCP) standards with independent monitoring. All adverse events and serious adverse events will be monitored and serious adverse events will be reported to Danish Medicines Agency.

ELIGIBILITY:
Inclusion Criteria:

* Admission with hypoxemic respiratory failure
* Age >= 18 years
* Expected duration of admission > 24 hours
* Need for oxygen supplementation to maintain SpO2 >= 88 % (patients at risk of hypercapnia) or SpO2 >= 94 % (other patients)
* Cognitively able to participate in the study
* Willing to participate and give informed consent

Exclusion Criteria:

* Need or anticipated need for mechanical ventilation (intermittent Continuous Positive Airway Pressure (CPAP) is allowed)
* Patients with CO-poisoning or other condition with unreliable SpO2.
* Patients in need of oxygen supplementation at more than 10 liters/min
* Pregnancy
* Cognitive or language barriers for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Probability of weaning from oxygen within 24 hours | 24 hours
  Fraction of patients weaned from oxygen supplementation within 24 hours

SECONDARY OUTCOMES:
Probability of weaning from oxygen within 12 hours | 12 hours
  Fraction of patients weaned from oxygen supplementation within 12 hours
Duration of admission | 30 days
  Time from admission to emergency department to discharge from hospital
Time within SpO2 target interval | 24 hours
  Fraction of time within prescribed SpO2 interval in O2matic and manual arm
Time with minor hypoxemia | 24 hours
  Fraction of time with SpO2 at 1 to 3 percentage points below target interval
Time with severe hypoxemia | 24 hours
  Fraction of time with SpO2 at 4 or more percentage points below target interval
Time with hyperoxia | 24 hours
  Fraction of time with SpO2 above target interval in O2matic and manual arm

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, DMSc, Study Chair — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Amager Hospital, Copenhagen
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Driscoll BR, Howard LS, Earis J, Mak V. British Thoracic Society Guideline for oxygen use in adults in healthcare and emergency settings. BMJ Open Respir Res. 2017 May 15;4(1):e000170. doi: 10.1136/bmjresp-2016-000170. eCollection 2017. No abstract available. PMID 28883921
- [Background] Cornet AD, Kooter AJ, Peters MJ, Smulders YM. The potential harm of oxygen therapy in medical emergencies. Crit Care. 2013 Apr 18;17(2):313. doi: 10.1186/cc12554. PMID 23635028
- [Background] Chu DK, Kim LH, Young PJ, Zamiri N, Almenawer SA, Jaeschke R, Szczeklik W, Schunemann HJ, Neary JD, Alhazzani W. Mortality and morbidity in acutely ill adults treated with liberal versus conservative oxygen therapy (IOTA): a systematic review and meta-analysis. Lancet. 2018 Apr 28;391(10131):1693-1705. doi: 10.1016/S0140-6736(18)30479-3. Epub 2018 Apr 26. PMID 29726345
- [Background] Hansen EF, Hove JD, Bech CS, Jensen JS, Kallemose T, Vestbo J. Automated oxygen control with O2matic(R) during admission with exacerbation of COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 14;13:3997-4003. doi: 10.2147/COPD.S183762. eCollection 2018. PMID 30587955